CLINICAL TRIAL: NCT06599645
Title: Impact of Combined Core Stability Training, Blood Flow Restriction, and Tai Chi on Muscle Physiology and Functional Characteristics Among Adults With Low Back Pain
Brief Title: Impact of Combined CST, BFR, and Tai Chi on Muscle Physiology and Functional Characteristics Among Adults With LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Lin Pipeng, Doctoral student, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LPipeng
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Tai Ji; Core stability; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): CST+BFR+Tai Chi+Education
  Interventions: Other: CST+BFR+Tai Chi+Education
- Group B (Experimental): CST+BFR+Education
  Interventions: Other: CST+BFR+Education
- Group C (Experimental): Tai Chi +BFR+Education
  Interventions: Other: Tai Chi +BFR+Education
- Group D (Other): CST+Education
  Interventions: Other: CST+Education

INTERVENTIONS:
Other: CST+BFR+Tai Chi+Education — 1. Core Stability Training: It includes core activation exercises (feed-forward control)(Libenson,2006). Each set will consist of 10 repetitions of this exercise with a 10-second hold. There will be a 30-second rest between repetitions and a 60-second rest after each set.
  2. Tai Chi: The first 10 Tai Chi movements from the 24-simplified Tai Chi form. Three qualified teachers will lead the training sessions.
  3. Blood Flow Restriction: The professional physical therapist puts on the cuff pneumatic tourniquet system(Kaastu Master) on the proximal end of the left lower limb of the subjects and gives a certain pressure through the Kaastu Master. The pressure needs to ensure that the venous return of the particapants is restricted to perfect ground, while the artery still has some blood flow.
  4. Education: After enrollment, patients will receive face-to-face education sessions at baseline, 30-45 min each time. Guided education by the same experienced professional physiotherapist.
  Arms: Group A
Other: CST+BFR+Education — 1. Core Stability Training: It includes core activation exercises (feed-forward control)(Libenson,2006). Each set will consist of 10 repetitions of this exercise with a 10-second hold. There will be a 30-second rest between repetitions and a 60-second rest after each set.
  2. Blood Flow Restriction: The professional physical therapist puts on the cuff pneumatic tourniquet system(Kaastu Master) on the proximal end of the left lower limb of the subjects and gives a certain pressure through the Kaastu Master. The pressure needs to ensure that the venous return of the particapants is restricted to perfect ground, while the artery still has some blood flow.
  3. Education: After enrollment, patients will receive face-to-face education sessions at baseline, 30-45 min each time. Guided education by the same experienced professional physiotherapist.
  Arms: Group B
Other: Tai Chi +BFR+Education — 1. Tai Chi: The first 10 Tai Chi movements from the 24-simplified Tai Chi form. Three qualified teachers will lead the training sessions.
  2. Blood Flow Restriction: The professional physical therapist puts on the cuff pneumatic tourniquet system(Kaastu Master) on the proximal end of the left lower limb of the subjects and gives a certain pressure through the Kaastu Master. The pressure needs to ensure that the venous return of the particapants is restricted to perfect ground, while the artery still has some blood flow.
  3. Education: After enrollment, patients will receive face-to-face education sessions at baseline, 30-45 min each time. Guided education by the same experienced professional physiotherapist.
  Arms: Group C
Other: CST+Education — 1. Core Stability Training: It includes core activation exercises (feed-forward control)(Libenson,2006). Each set will consist of 10 repetitions of this exercise with a 10-second hold. There will be a 30-second rest between repetitions and a 60-second rest after each set.
  2. Education: After enrollment, patients will receive face-to-face education sessions at baseline, 30-45 min each time. Guided education by the same experienced professional physiotherapist.
  Arms: Group D

SUMMARY:
Background:

Low back pain (LBP) is highly prevalent globally, affecting people of all ages(Wu et al., 2020). In China, LBP is a leading cause of disease burden(Wu et al., 2019). Exercise therapy such as core stability training(CST), Tai Chi(TC) and education are commonly recommended treatments, but research on optimal protocols has been limited. Blood flow restriction(BFR) is beneficial for inducing muscle hypertrophy and promoting muscle strength (Hughes et al., 2019). Combined approaches using multiple modalities may provide added benefits but are understudied.

Research objectives:

1. To determine the effects of combined CST, BFR and Tai Chi on muscle physiology (muscle activation, muscle fatigue, back extensor strength, and transverses abdominus control) among working adults with LBP.
2. To determine the effects of combined CST+ BFR+Tai Chi on functional performance (gait speed, balance, proprioception, and postural sway) among working adults with LBP.
3. To determine the effects of combined CST+BFR+Tai Chi on pain intensity among working adults with LBP.
4. To determine the effects of combined CST+BFR+Tai Chi on fear among working adults with LBP.

Location of research:

Qianxinan Wutong Orthopedic Hospital, Guizhou Province, China

Instrumentations:

1. Demographic Data
2. Surface Electromyography (S-EMG)
3. Pressure Biofeedback Unit (PBU)
4. Back Extensor Strength Test (BEST)
5. Joint Repositioning Error(JRE)
6. APECS app
7. Y-Balance Test(YBT)

8.10-Meter Walk Test(10MWT)

9.Visual Analogue Scale (VAS)

10.Chinese version of the Fear-Avoidance Beliefs Questionnaire(FABQ-CHI)

Interventions:

Group A: CST+BFR+Tai Chi+Education;

Group B: CST+BFR+Education;

Group C: Tai Chi +BFR+Education;

Group D: CST+Education.

Sample size:

Considering 30% drop out. 52 participants. 13 participants in each group

Statistical analysis:

Data were processed using SPSS version 25.0 and Microsoft Excel 2010 software.

1. Demographic data = descriptive analytics.
2. All objectives = repeated measure ANCOVA (within-between interactions) for all variables.
3. The significant level is P < 0.05.

DETAILED DESCRIPTION:
Research objectives:

1. To determine the effects of combined CST, BFR and Tai Chi on muscle physiology (muscle activation, muscle fatigue, back extensor strength, and transverses abdominus control) among working adults with LBP.
2. To determine the effects of combined CST+ BFR+Tai Chi on functional performance (gait speed, balance, proprioception, and postural sway) among working adults with LBP.
3. To determine the effects of combined CST+BFR+Tai Chi on pain intensity among working adults with LBP.
4. To determine the effects of combined CST+BFR+Tai Chi on fear among working adults with LBP.

Test methods for each indicator:

1. The RMS and MF value test by S-EMG

   For each muscle, double electrode sheets are put to the belly. The electrode placement site is as follows: ①Erecter spinae: Open 2cm lateral to the midline of the trunk, between the spinous process of the twelfth thoracic vertebra and the first lumbar vertebra. ②Multifidus: 2cm next to the L4-5 interspinous. ③Rectus abdominis: On both sides of the midline of the abdomen, 3cm away from the navel. ④Transversus abdominis: Approximately 2 cm medial to the intersection of the vertical line traversing the anterior superior iliac spine and the lower border of the costal arch.

   Test action: Back Bridge, Side Bridge, Abdominal Bridge. Each action lasts 10 seconds, and there is a 2-minute break between two adjacent actions to ensure that muscle weariness from the previous measurement does not interfere with the following measurement.

   S-EMG analysis: It is the recording of electrical activity in muscles utilizing the BioForce surface electromyography tester model JE-TB1610 and the accompanying wireless data collection equipment. The sampling frequency was 2000Hz, the above three exercise groups lasted 10 seconds each, and the original EMG signal was recorded for 10 seconds. Use the InstallShield Wizard operating software to execute 10-500Hz noise processing on the original muscle electrical data(Perchthaler et al., 2015). Then, from the 3rd to the 7th second, extract the data, remove the baseline, demodulate and smooth the original signal, take the absolute value of the signal during the demodulation process, and acquire the average value of the EMG data from the 3rd to the 7th second (RMS value, MF value).
2. Transverses abdominus control test

   In the case of muscle control, which is quantified by PBU. In the prone position, the transversus abdominis will be tested. The inflated cuff will be placed beneath the abdomen at the anterior superior iliac spine level. The patient will be asked to draw in the lower abdomen without moving the upper stomach, back, or pelvis once the PBU has been inflated to 70 mm Hg. Readings will be taken at the end of a 10-second contraction. Two submaximal force tests will be performed to familiarise participants with each test position, followed by two repeats of maximum isometric contraction. For analysis, the average of the two greatest contractions will be used(Cairns et al., 2000).
3. Back extensor strength test

   The participant will be seated on the treatment table with their head in the midline, trunk straight, arms along their body, palms facing upwards, and feet over the table's edge. The dynamometer will be placed at the inferior angle of the scapulae, in the center of the back between the shoulder blades. The therapist will be above and to the side of the patient. The test will be executed by the guidelines of Yang et al. (2020). After obtaining the proper starting posture, the participant will be asked to relax their arms, lift their head and chest, and push back against the dynamometer for 5 seconds with maximal force (N) .
4. Lumbar proprioception test

   The procedure utilized for the proprioception test was reported by Puntumetakul(2018). "The participant was seated (90° hips and knees) with feet on the ground and hands on thighs, and the examiner guided the participant into the neutral lumbar spine position." The center of the 10-centimeter tape measure was placed on sacral segment 1 (S1) as the measurement's starting point. The start point was marked by a laser pointer with a stable foundation. The examiner advised the participant to "remember the target position, then perform the maximum anterior and posterior pelvic tilt twice, holding each position for five seconds," before returning to the neutral target position. As a combined repositioning error, deviation from the starting location was assessed in centimeters. The participant received no feedback regarding any errors. The participants practiced the relocation test twice before the evaluation. This examination process was repeated three times with one-minute rest intervals in between. For analysis, the mean values will be employed.
5. Trunk postural sway test

   According to Trovato et al.(2020), APECS will record the participants in a standing stance for the 30s, and participants will be asked to wear little clothes to reduce biases associated with incorrect landmark positioning during the postural analysis; for the same reason, trained clinicians will place markers on the participants' bodies in correlation to the app's specified landmarks. One video will be taken for the sagittal plane (left). Participants will be told to keep their feet the same width as their shoulders. Finally, the videos that meet the regulations will be imported into the video analysis system in APECS for analysis. The maximum angle of the torso wobbles will be recorded and used for analysis.
6. Standing dynamic balance test

   While standing on one leg (barefoot) in a central location on the Y-Balance Test instrument, with hands on the wing of the ilium, the subjects will be asked to move the pointer as far as possible in three directions - anterior, posteromedial, and posterolateral. All Y-Balance Test efforts will be made in the same order: first in the anterior direction, then in the posterolateral direction, and finally in the posteromedial direction. Participants moved the pointer with their dominant leg first. The following is the measuring protocol (Linek et al., 2017): 1. A training effort consists of four replications of the right and left lower limbs in each of three directions: anterior, posteromedial, and posterolateral. 2. Execution of the proper test, which consisted of three attempts in each direction, measuring the distance between the pointer's closest location and the central plate. Only when the individual tested was able to return to the starting location while fully controlling the movement was the result of each attempt saved. During the performance of an attempt, the following will be considered irregularities: support using the movement-performing limb on the surface of the pointer to maintain balance, pushing the pointer to achieve a better result, changing the starting position (taking the upper limbs off the iliac wing). In such a case, the participant repeated the attempt until three properly accomplished repetitions were obtained (Linek et al., 2017). For the analysis, the maximum reach distance in each direction and the composite score are employed (Picot et al., 2021)
7. Gait speed test

   For gait speed, a 10-meter walk test was used, which required the participant to walk for 10 meters in a straight line at their normal speed, with a 1-meter start-up before starting timing and a 1-meter stop-time timing. It is permissible to employ an assistance walking device. For the walking test, each participant completed three consecutive trials. The participants are told to "walk at your normal, comfortable pace" until they reach the end of the indicated course. The duration is recorded using a stopwatch, which is started when the participant's lead leg (or assistive device) crosses the first marker and stopped when the participant's lead leg (or assistive device) crosses the second marker. By dividing the distance of 8 m by the time recorded, the recorded time is translated into walking speed (m/s).
8. Fear avoidance belief test

   The subject will next be allowed 3-5 minutes to respond to the FABQ-CHI. Those who are unable to read will receive assistance.
9. Pain test

Finally, the subject will be allowed 2-3 minutes to respond to the VAS. The following is the specific evaluation method: Choose a 10 cm ruler and face the experimenter with it marked with a complete digital scale from 0 to 10. The patient only sees scales at both ends of the ruler, and the 0 end is blank. "No pain" implies no pain at all, "14" means mild pain, "56" means moderate discomfort, "7" or more means severe pain, and "10" signifies agonizing pain(Langley & Sheppard, 1985). When the low back pain arises on the 0 scale, the patient begins to picture his pain state, and the experimenter notes the ultimate number, which can be immediately recorded as the patient's pain intensity score(Wewers & Lowe, 1990).

Rest for 30-60 seconds between tests to remove the confounding impact of weariness.

Procedure

This study will screen subjects according to inclusion and exclusion criteria. Before the evaluation and examination, the physiotherapist will tell the participants the purpose and methods, and the participants need to sign the consent form. The demographic data, which includes biographical information, short questions concerning the occurrence of LBP, and past medical history, will then be recorded. The subjects must then complete the anthropometric data, such as weight, height, and BMI. All patients require blood pressure and heart rate measurements before and after treatment.

For all subjects, the measurement indicators will be measured before the intervention, six weeks after the treatment, and 12 weeks after the treatment. In addition, all the subjects need to perform a warm-up before each exercise intervention and a cooldown after the exercise intervention. Warm up includes walking (5 min) and dynamic stretching (5 mins). Cooldown includes static stretching (5 min).

For group A, subjects will receive education from a qualified physiotherapist before the first treatment. Subsequent treatment begins with a warm-up. After the warm up, the physical therapist will install the BFR device for the subject as required. Then, the patients will receive CST for 15 minutes. Then, they will receive Tai Chi practice for 15 minutes. Finally, complete a 5-minute cooldown. The above treatments are performed 3 times a week for 12 weeks(Zou, Zhang, Liu, et al., 2019).

For group B, subjects will receive education from a qualified physiotherapist before the first treatment. Subsequent treatment begins with a warm-up. After the warm up, the physical therapist will install the BFR device for the subject as required. Then, the patients will receive CST for 30 minutes. Finally, complete a 5-minute cooldown. The above treatments are performed 3 times a week for 12 weeks(Nipa et al., 2022).

For group C, subjects will receive education from a qualified physiotherapist before the first treatment. Subsequent treatment begins with a warm-up. After the warm up, the physical therapist will install the BFR device for the subject as required. Then, the patients will receive Tai Chi for 30 minutes. Finally, complete a 5-minute cooldown. The above treatments are performed 3 times a week for 12 weeks(Qin et al., 2019).

For group D, subjects will receive education from a qualified physiotherapist before the first treatment. Subsequent treatment begins with a warm-up. Then, the patients will receive CST for 30 minutes. Finally, complete a 5-minute cooldown. The above treatments are performed 3 times a week for 12 weeks(Nipa et al., 2022).

Statistical analysis:

Data were processed using SPSS version 25.0 and Microsoft Excel 2010 software.

1. Demographic data = descriptive analytics.
2. All objectives = repeated measure ANCOVA (within-between interactions) for all variables.
3. The significant level is P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All participants had stable vital signs, were cognizant, and had no cognitive impairment.
* Aged 18-60 years old, able to understand Mandarin Chinese, and willing to cooperate.
* LBP duration ≥ 3 months.
* Be diagnosed as NLBP.
* VAS score ≤ 5 points.

Exclusion Criteria:

* Patients with severe heart disease, liver disease, renal disease, pulmonary insufficiency, tumors, and postoperative dysfunction.
* Patients who are unconscious and unable to cooperate.
* Spinal fractures, severe arthritis, bony spinal stenosis, ankylosing spondylitis, open fractures, or unhealed traumatic wounds.
* Patients who have not been diagnosed with NLBP.
* Unable to communicate and read in Chinese.
* Age <18 & >60 years old.
* LBP duration < 3 months.
* Patients with high blood pressure and abnormal heartbeat.
* VAS score > 5 points.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Core muscle activation by root mean square(RMS) | Baseline (1st week), 6th week, and 12th week
  Root Mean Square (RMS) is a vector used to analyze the properties of electrical signal fluctuations, and the size of the RMS value represents the level of activity of a certain muscle(Abdelouahad et al., 2018). Absolute RMS demonstrated the highest overall dependability (ICC: 0.66-0.98) across activities (ICC: 0.66-0.98)(Van Helden et al., 2022).
Core muscle fatigue by mean frequency (MF) | Baseline (1st week), 6th week, and 12th week
  Mean Frequency (MF) is a frequency-domain index that represents the midpoint of muscle fiber discharge frequency during skeletal muscle contraction. It is widely assumed that it is connected to the proportion of fast and slow fibers in muscle tissue. The multifidus muscle demonstrated good to outstanding reproducibility of initial MF and MF fatigue changes during Trunk Holding Tests (ICCwithindays =82%; ICCbetweendays =78%) (Ng & Richardson, 1996).
Abdominal drawing-in maneuver by the pressure biofeedback unit (PBU) | Baseline (1st week), 6th week, and 12th week
  The Pressure Biofeedback Unit (PBU) device consists of a pressure transducer with three airbags, a catheter, and a sphygmomanometer (with a range of 0 to 200 mmHg). It will be applied to evaluate abdominal drawing-in movements objectively (Grooms et al., 2013b). It is a trustworthy clinical instrument for assessing deep abdominal muscle function, with moderate to good (ICC = 0.47-0.82) and acceptable construct validity (ICC = 0.48-0.90) (P. O. D. P. Lima et al., 2011).
Back Extensor Strength by a push-pull dynamometer | Baseline (1st week), 6th week, and 12th week
  A push-pull dynamometer will be applied to assess back extensor strength in the prone position. Because of its acceptable reliability (ICC=0.93), validity (r=0.54), and measurement errors, maximal isometric back extensor strength assessment in a prone posture can be applied to individuals with varying levels of back strength and may be the most useful for ranking back extensor strength in clinical and epidemiological studies (Yang et al., 2020).
Postural sway by the mobile app APECS | Baseline (1st week), 6th week, and 12th week
  The application of a mobile app could represent a quick, safe, and accurate method for researchers and clinicians to evaluate general posture quantitatively. Adopting a movable and affordable tool for postural assessment could benefit the primary prevention of musculoskeletal disorders of the spine. The mobile app APECS-AI Posture Evaluation and Correction System® (New Body Technologies SAS, Grenoble, France) (APECS app) will be applied to evaluate the subject's postural sway in this study. The evaluation index is the maximum angle of the torso wobbles. According to a recommendation from a study, clinicians should consider APECS's worth as an auxiliary posture evaluation tool with (ICC > 0.60) (Trovato et al., 2022).
Balance by Y-Balance Test | Baseline (1st week), 6th week, and 12th week
  The Y-Balance Test Kit will be applied to measure balance in this study. The device includes a single central plastic plate and three attached tubes positioned anteriorly, posteromedially, and posterolaterally. A measurement with a 0.5 cm spacing is placed on each of the tubes. A study found that the Y-Balance Test has high inter-rater reliability and validity for assessing dynamic balance in the CLBP group (Alshehre et al., 2021).
Lumbar proprioception by joint repositioning error(JRE) | Baseline (1st week), 6th week, and 12th week
  The primary result of proprioception was a joint repositioning error(JRE). The absolute error, constant error, and variable error can all be used to describe repositioning errors. We picked absolute error since it affects accuracy(Strimpakos et al., 2006), reflects the magnitude of the inaccuracy (Sheeran et al., 2012), and is the most widely used measurement (Tong et al., 2017). The proprioception test had great inter-rater reliability(ICC=0.61-0.76)(Petersen & Rundquist, 2009).
Gait speed by the 10-meter walk test. | Baseline (1st week), 6th week, and 12th week
  The gait speed is measured using the 10-Meter Walk Test. The gait speed test is the most commonly used outcome measure to assess functional limitations of the lower limbs (Muñoz-Mendoza et al., n.d.). With ICC values ranging from 0.96 to 0.98, 10m gait speed measurement shows outstanding test-retest reliability(Peters et al., 2013).
Fear avoidance belief by the Chinese version of the Fear-avoidance Beliefs. Questionnaire (FABQ-CHI) | Baseline (1st week), 6th week, and 12th week
  The Chinese version of the Fear-avoidance Beliefs Questionnaire (FABQ-CHI) is a relatively basic, easy-to-understand, easy-to-use, low-cost, and comprehensive LBP evaluation tool. The FABQ-CHI was shown to have adequate factor structure, internal consistency, test-retest reliability, and construct validity. (Pei et al., 2010). The maximum possible score for each question is 6, the lowest possible score is 0, and the total score is 96. The higher the score, the greater the severity of the perceived fear-avoidance belief.
Pain by visual analogue scale (VAS) | Baseline (1st week), 6th week, and 12th week
  Visual Analogue Scale (VAS) is a 10 cm horizontal strip with numbers ranging from 0 to 10 (the most severe pain possible). This is one of the most dependable quantitative scales that is commonly utilized in research (Scrimshaw & Maher, 2001). VAS has proven to be trustworthy and valid (ICC=0.49-0.83) (Crossley et al., 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Zarina Zahari, Doctor, Study Director — Centre of Physiotherapy, Faculty of Health Sciences, Universiti Teknologi MARA, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelraouf OR, Abdel-Aziem AA. THE RELATIONSHIP BETWEEN CORE ENDURANCE AND BACK DYSFUNCTION IN COLLEGIATE MALE ATHLETES WITH AND WITHOUT NONSPECIFIC LOW BACK PAIN. Int J Sports Phys Ther. 2016 Jun;11(3):337-44. PMID 27274419
- [Background] Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol (1985). 2006 May;100(5):1460-6. doi: 10.1152/japplphysiol.01267.2005. Epub 2005 Dec 8. PMID 16339340
- [Background] Ainpradub K, Sitthipornvorakul E, Janwantanakul P, van der Beek AJ. Effect of education on non-specific neck and low back pain: A meta-analysis of randomized controlled trials. Man Ther. 2016 Apr;22:31-41. doi: 10.1016/j.math.2015.10.012. Epub 2015 Nov 2. PMID 26585295
- [Background] Dos Santos LP, Santo RCDE, Ramis TR, Portes JKS, Chakr RMDS, Xavier RM. The effects of resistance training with blood flow restriction on muscle strength, muscle hypertrophy and functionality in patients with osteoarthritis and rheumatoid arthritis: A systematic review with meta-analysis. PLoS One. 2021 Nov 10;16(11):e0259574. doi: 10.1371/journal.pone.0259574. eCollection 2021. PMID 34758045
- [Background] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Background] Hughes L, Rosenblatt B, Haddad F, Gissane C, McCarthy D, Clarke T, Ferris G, Dawes J, Paton B, Patterson SD. Comparing the Effectiveness of Blood Flow Restriction and Traditional Heavy Load Resistance Training in the Post-Surgery Rehabilitation of Anterior Cruciate Ligament Reconstruction Patients: A UK National Health Service Randomised Controlled Trial. Sports Med. 2019 Nov;49(11):1787-1805. doi: 10.1007/s40279-019-01137-2. PMID 31301034
- [Background] Korakakis V, Whiteley R, Epameinontidis K. Blood Flow Restriction induces hypoalgesia in recreationally active adult male anterior knee pain patients allowing therapeutic exercise loading. Phys Ther Sport. 2018 Jul;32:235-243. doi: 10.1016/j.ptsp.2018.05.021. Epub 2018 May 31. PMID 29879638
- [Background] Paungmali A, Henry LJ, Sitilertpisan P, Pirunsan U, Uthaikhup S. Improvements in tissue blood flow and lumbopelvic stability after lumbopelvic core stabilization training in patients with chronic non-specific low back pain. J Phys Ther Sci. 2016 Jan;28(2):635-40. doi: 10.1589/jpts.28.635. Epub 2016 Feb 29. PMID 27064327
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Qin J, Zhang Y, Wu L, He Z, Huang J, Tao J, Chen L. Effect of Tai Chi alone or as additional therapy on low back pain: Systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Sep;98(37):e17099. doi: 10.1097/MD.0000000000017099. PMID 31517838
- [Background] Semeru GM, Halim MS. Acceptance versus catastrophizing in predicting quality of life in patients with chronic low back pain. Korean J Pain. 2019 Jan;32(1):22-29. doi: 10.3344/kjp.2019.32.1.22. Epub 2019 Jan 2. PMID 30671200
- [Background] Smith BE, Littlewood C, May S. An update of stabilisation exercises for low back pain: a systematic review with meta-analysis. BMC Musculoskelet Disord. 2014 Dec 9;15:416. doi: 10.1186/1471-2474-15-416. PMID 25488399
- [Background] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064
- [Background] Wang R, Zhu D, Wang L, Liu J, Zou J, Sun Y, Jiang Y, Hu HY, Deng ZW, Weng LM, Zheng KY, Kiartivich S, Wang XQ. Tai Chi Quan Versus Physical Therapy on Pain and Cognitive Performance for Elderly People With Chronic Low Back Pain: Study Protocol for a Randomized Controlled Trial. Front Aging Neurosci. 2022 Jun 16;14:900430. doi: 10.3389/fnagi.2022.900430. eCollection 2022. PMID 35783144
- [Background] Wang XQ, Xiong HY, Du SH, Yang QH, Hu L. The effect and mechanism of traditional Chinese exercise for chronic low back pain in middle-aged and elderly patients: A systematic review. Front Aging Neurosci. 2022 Oct 10;14:935925. doi: 10.3389/fnagi.2022.935925. eCollection 2022. PMID 36299610
- [Background] Wu A, Dong W, Liu S, Cheung JPY, Kwan KYH, Zeng X, Zhang K, Sun Z, Wang X, Cheung KMC, Zhou M, Zhao J. The prevalence and years lived with disability caused by low back pain in China, 1990 to 2016: findings from the global burden of disease study 2016. Pain. 2019 Jan;160(1):237-245. doi: 10.1097/j.pain.0000000000001396. PMID 30234697
- [Background] Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Transl Med. 2020 Mar;8(6):299. doi: 10.21037/atm.2020.02.175. PMID 32355743
- [Background] Yue YS, Wang XD, Xie B, Li ZH, Chen BL, Wang XQ, Zhu Y. Sling exercise for chronic low back pain: a systematic review and meta-analysis. PLoS One. 2014 Jun 11;9(6):e99307. doi: 10.1371/journal.pone.0099307. eCollection 2014. PMID 24919119